CLINICAL TRIAL: NCT06522711
Title: Virtual Reality as a Strategy for Intra-operatory Anxiolysis and Pharmacological Sparing in Patients Undergoing Breast Surgeries : the V-RAPS Randomized Controlled Trial
Brief Title: Virtual Reality for Anxiolysis and Pharmacological Sparing
Acronym: V-RAPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Paperplane Therapeutics (Unknown)
Responsible Party: Principal Investigator, Pascal Laferrière-Langlois, Clinical assistant professor, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-3802
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Virtual Reality; Propofol
Keywords: Virtual reality; Anxiety; Patient-controlled sedation; Pain; Propofol; Breast surgery
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: After the participants meet all the inclusion criteria and meet no exclusion criteria, patients will then be randomized by an unbiased algorithm in a 1 for 1 ratio (one control patient for each patient in the virtual reality group). However, the chosen scenario in the virtual reality group will be a result of each patient's personal preference; the patients will also be able to switch between scenarios at will.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual reality (Experimental): Patients assigned to use a virtual reality headset during their surgery.
  Interventions: Device: Virtual reality headset
- Control (Active Comparator): Standard of care group.
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: Virtual reality headset — A brief overview of all three virtual reality scenarios will be shown in a consolidated video prior to letting the participant select the preferred scenario. The participant's choice of scenario will then be documented. Once paravertebral blocks are completed and the participants are in supine position and the surgeon is ready to disinfect, the VR headset will be applied on the face of the participants in the intervention group and the chosen scenario will be started. If at any point the patient expresses a desire to stop using VR during the surgery, we will first offer them an alternate scenario. If they reiterate their willingness to stop, with or without having experienced the new scenario, the headset will be removed for the remainder of the surgery.
  Arms: Virtual reality
Other: Standard of care — Standard of care in anesthesia with patient-controlled sedation.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn if virtual reality can reduce propofol requirements in adult, female patients undergoing elective breast surgery under regional anesthesia. The main question it aims to answer is:

Can virtual reality immersion reduce intra-operative propofol requirements in adult female patients undergoing elective breast surgery under regional anesthesia?

Researchers will compare time and weight-adjusted average propofol requirements in both the intervention group and the control group to see if there is a reduction in sedative usage in the group using the virtual reality device.

Participants will be randomly assigned to either a virtual reality (intervention) group or a control group.

* The patients in the virtual reality group will have a virtual reality headset on during the surgery with a preselected scenario of their choice.
* Both groups will have access to patient-controlled sedation under the supervision of an anesthesiologist and will be permitted to self-administer propofol boluses as needed.

DETAILED DESCRIPTION:
Virtual reality (VR) has carved out a growing place for itself in our leisure activities, video games and even in medicine. Recent studies show that VR can reduce anxiety and pain in patients undergoing uncomfortable care (e.g. wound care, dental care, venous access). While the population most frequently investigated is pediatric, the benefits can be extended to other populations. The operating room is uncommon due to the type of procedure and the older patient profile. Yet, with the democratization of regional and neuraxial anesthesia, VR could improve the patient experience in the operating room.

The main objective of this study is to explore the impact of VR on intravenous (I.V.) sedation requirements in adult patients undergoing breast surgery under paravertebral (PV) block. The hypothesis is that VR will serve as an effective distraction in the operative context, reducing the need for pharmacology. In parallel, multiple secondary objectives will also be explored, such as the evaluation of the tolerance to the VR headset, the impact of the chosen type of scenario on the primary outcome, the incidence of adverse effects, the variation of the Nociception Level Index (NOL index) in awake patients as well as overall patient satisfaction.

This single center, open-label, randomized controlled trial will be conducted in a Canadian academic hospital. 100 patients above the age of 18 years undergoing breast surgery (mastectomy, reduction, augmentation, reconstruction, etc.) under regional anesthesia, specifically paravertebral block, will be included in this study. Patients will be randomized either to the intervention group or the control group. The intervention group will have a VR helmet and the control group a standard treatment. Both will have access to patient-controlled sedation (PCS), self-administering their own sedation under clinical observation. Patients in the VR group will be able to choose, before the procedure begins, between 3 different VR environments and will also be allowed to switch between these environments during the surgery. The primary outcome of this study will be the time-weighted dose of propofol (sedative) self-administered during the procedure. Secondary outcomes will include patient satisfaction, premature removal of VR helmet, presence of nausea, desaturation, hypotension and post-anesthesia monitoring time.

ELIGIBILITY:
Inclusion Criteria:

* Fully consented female patients above the age of 18 years;
* Undergoing elective, awake, breast surgery performed under paravertebral block.

Exclusion Criteria:

* Hearing or visual impairment;
* History of epilepsy, seizure or severe dizziness;
* Severe mental impairment;
* Recent eye or facial surgery or wounds;
* Inability to use the VR hand controller.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Propofol self-administration | Between 1 hour and 3 hours
  Time-adjusted and weight-adjusted average self-administration of propofol in mcg/kg/min in female patients undergoing breast surgery under paravertebral block.

SECONDARY OUTCOMES:
Preoperative anxiety | Up to 1 hour
  Level of anxiety before the surgery evaluated by the Amsterdam Preoperative Anxiety and Information Scale.
Remifentanil administration | Between 1 hour and 3 hours
  Time-adjusted and weight-adjusted average administration of remifentanil in mcg/kg/min.
Ketamine administration | Between 1 hour and 3 hours
  Weight-adjusted administration of ketamine in mg/kg.
Adverse events | Between 1 hour and 3 hours
  The incidence of adverse events such as cybersickness, nausea, bradycardia, desaturation and hypotension.
Scenario switches | Between 1 hour and 3 hours
  Percentage of patients that switched scenarios.
Virtual reality usage | Between 1 hour and 3 hours
  The total time, in minutes, as well as the relative time compared to the duration of the surgery, expressed as a percentage, during which the VR headset was worn.
Virtual reality usage per first scenario | Between 1 hour and 3 hours
  Total duration in minutes spent by the patient on the VR scenario chosen, and the order in which VR scenarios were presented.
Virtual reality headset removal | Between 1 hour and 3 hours
  Percentage of patients that removed the headset before the end of the surgery.
Post-Anesthesia Care Unit stay | Between 30 minutes and 2 hours
  The total time in minutes spent in the PACU.
Enthusiasm at the idea of using virtual reality | Up to 1 hour
  Initial enthusiasm at the idea of using a VR headset during surgery assessed on a 10 point Likert scale.
Ease of use | Between 30 minutes and 2 hours
  Ease of use of the virtual reality technology assessed on a 10 point Likert scale.
Enjoyment of the first scenario chosen | Between 30 minutes and 2 hours
  Enjoyment of the first scenario chosen assessed on a 10 point Likert scale.
Overall satisfaction | Between 30 minutes and 2 hours
  Overall satisfaction with the experience assessed on a 10 point Likert scale
NOL index readings | Between 1 hour and 3 hours
  NOL index readings over time per patient, assessed continuously.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Laferriere-Langlois, MD, MSc, Principal Investigator — Ciusss de L'Est de l'Île de Montréal
Locations (1):
- Maisonneuve-Rosemont Hospital - CIUSSS de l'Est de l'Île de Montréal, Montreal East, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boutin J, Kamoonpuri J, Faieghi R, Chung J, de Ribaupierre S, Eagleson R. Smart haptic gloves for virtual reality surgery simulation: a pilot study on external ventricular drain training. Front Robot AI. 2024 Jan 10;10:1273631. doi: 10.3389/frobt.2023.1273631. eCollection 2023. PMID 38269073
- [Background] Boyce L, Jordan C, Egan T, Sivaprakasam R. Can virtual reality enhance the patient experience during awake invasive procedures? A systematic review of randomized controlled trials. Pain. 2024 Apr 1;165(4):741-752. doi: 10.1097/j.pain.0000000000003086. Epub 2023 Oct 23. PMID 37870233
- [Background] Eijlers R, Utens EMWJ, Staals LM, de Nijs PFA, Berghmans JM, Wijnen RMH, Hillegers MHJ, Dierckx B, Legerstee JS. Systematic Review and Meta-analysis of Virtual Reality in Pediatrics: Effects on Pain and Anxiety. Anesth Analg. 2019 Nov;129(5):1344-1353. doi: 10.1213/ANE.0000000000004165. PMID 31136330
- [Background] Fuica R, Krochek C, Weissbrod R, Greenman D, Freundlich A, Gozal Y. Reduced postoperative pain in patients receiving nociception monitor guided analgesia during elective major abdominal surgery: a randomized, controlled trial. J Clin Monit Comput. 2023 Apr;37(2):481-491. doi: 10.1007/s10877-022-00906-1. Epub 2022 Aug 17. PMID 35976578
- [Background] Gelinas C, Shahiri T S, Richard-Lalonde M, Laporta D, Morin JF, Boitor M, Ferland CE, Bourgault P, Richebe P. Exploration of a Multi-Parameter Technology for Pain Assessment in Postoperative Patients After Cardiac Surgery in the Intensive Care Unit: The Nociception Level Index (NOL)TM. J Pain Res. 2021 Dec 7;14:3723-3731. doi: 10.2147/JPR.S332845. eCollection 2021. PMID 34908872
- [Background] Hitching R, Hoffman HG, Garcia-Palacios A, Adamson MM, Madrigal E, Alhalabi W, Alhudali A, Sampaio M, Peterson B, Fontenot MR, Mason KP. The Emerging Role of Virtual Reality as an Adjunct to Procedural Sedation and Anesthesia: A Narrative Review. J Clin Med. 2023 Jan 20;12(3):843. doi: 10.3390/jcm12030843. PMID 36769490
- [Background] Huang MY, Scharf S, Chan PY. Effects of immersive virtual reality therapy on intravenous patient-controlled sedation during orthopaedic surgery under regional anesthesia: A randomized controlled trial. PLoS One. 2020 Feb 24;15(2):e0229320. doi: 10.1371/journal.pone.0229320. eCollection 2020. PMID 32092098
- [Background] Kreienbuhl L, Elia N, Pfeil-Beun E, Walder B, Tramer MR. Patient-Controlled Versus Clinician-Controlled Sedation With Propofol: Systematic Review and Meta-analysis With Trial Sequential Analyses. Anesth Analg. 2018 Oct;127(4):873-880. doi: 10.1213/ANE.0000000000003361. PMID 29750696
- [Background] Kuhn AW, Yu JK, Gerull KM, Silverman RM, Aleem AW. Virtual Reality and Surgical Simulation Training for Orthopaedic Surgery Residents: A Qualitative Assessment of Trainee Perspectives. JB JS Open Access. 2024 Mar 20;9(1):e23.00142. doi: 10.2106/JBJS.OA.23.00142. eCollection 2024 Jan-Mar. PMID 38511201
- [Background] Lu Y, Hao LX, Chen L, Jin Z, Gong B. Systematic review and meta-analysis of patient-controlled sedation versus intravenous sedation for colonoscopy. Int J Clin Exp Med. 2015 Nov 15;8(11):19793-803. eCollection 2015. PMID 26884890
- [Background] Rudkin GE, Osborne GA, Curtis NJ. Intra-operative patient-controlled sedation. Anaesthesia. 1991 Feb;46(2):90-2. doi: 10.1111/j.1365-2044.1991.tb09345.x. PMID 1872456
- [Background] Ryu S, Kitagawa T, Goto K, Okamoto A, Marukuchi R, Hara K, Ito R, Nakabayashi Y. Intraoperative Holographic Guidance Using Virtual Reality and Mixed Reality Technology During Laparoscopic Colorectal Cancer Surgery. Anticancer Res. 2022 Oct;42(10):4849-4856. doi: 10.21873/anticanres.15990. PMID 36192000
- [Background] Wang Y, Guo L, Xiong X. Effects of Virtual Reality-Based Distraction of Pain, Fear, and Anxiety During Needle-Related Procedures in Children and Adolescents. Front Psychol. 2022 Apr 19;13:842847. doi: 10.3389/fpsyg.2022.842847. eCollection 2022. PMID 35519646
- [Background] Yamashita Y, Aijima R, Danjo A. Clinical effects of different virtual reality presentation content on anxiety and pain: a randomized controlled trial. Sci Rep. 2023 Nov 22;13(1):20487. doi: 10.1038/s41598-023-47764-8. PMID 37993645
- [Background] Yi WS, Rouhi AD, Duffy CC, Ghanem YK, Williams NN, Dumon KR. A Systematic Review of Immersive Virtual Reality for Nontechnical Skills Training in Surgery. J Surg Educ. 2024 Jan;81(1):25-36. doi: 10.1016/j.jsurg.2023.11.012. Epub 2023 Nov 30. PMID 38036388
- [Derived] Zako J, Daccache N, Burey J, Clairoux A, Morisson L, Laferriere-Langlois P. Virtual reality as a strategy for intra-operatory anxiolysis and pharmacological sparing in patients undergoing breast surgeries: The V-RAPS randomized controlled trial protocol. PLoS One. 2025 Jul 7;20(7):e0327555. doi: 10.1371/journal.pone.0327555. eCollection 2025. PMID 40622954